CLINICAL TRIAL: NCT00350636
Title: Multi-Center, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Daily Dosing With Oxybutynin Topical Gel to Treat the Symptoms of Overactive Bladder With a 14-Week Open-Label Safety Extension
Brief Title: A Comparison of a New Drug to Treat Overactive Bladder vs. Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel PhD, Executive Director, Watson
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OG05009
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-04

CONDITIONS: Overactive Bladder
Keywords: OAB, anticholineric, oxybutynin, urge urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin topical gel (Experimental): Oxybutynin topical gel
  Interventions: Drug: Oxybutynin topical gel
- Placebo topical gel (Placebo Comparator): placebo topical gel
  Interventions: Other: Placebo topical gel

INTERVENTIONS:
Drug: Oxybutynin topical gel — 1 application daily to skin for 12 weeks
  Other Names: Oxybutynin
  Arms: Oxybutynin topical gel
Other: Placebo topical gel — 1 application daily to skin for 12 weeks
  Other Names: Placebo
  Arms: Placebo topical gel

SUMMARY:
A new drug for overactive bladder is compared to placebo to determine if it is safe and effective. The study lasts approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females and males, 18 years of older with overactive bladder symptoms

Exclusion Criteria:

* Treatable conditions that may cause urinary incontinence
* Medical conditions in which it would be unsafe to use an anti-cholinergic agent.
* The use of concomitant drugs that would confound the efficacy evaluation.
* The use of concomitant drugs that would be unsafe with an anti-cholinergic agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Caramelli, MS, Study Director — Watson Pharmaceuticals
Locations (63):
- United States (63):
  - Birmingham, Alabama
  - Homewood, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Buena Park, California
  - Laguna Woods, California
  - Sacramento, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Waterbury, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Leesburg, Florida
  - Ocala, Florida
  - Plantation, Florida
  - Tallahassee, Florida
  - West Palm Beach, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Belville, Illinois
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Shreveport, Louisiana
  - Watertown, Massachusetts
  - Saginaw, Michigan
  - Saint Joseph, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Albany, New York
  - Garden City, New York
  - New York, New York
  - Williamsville, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Bethany, Oklahoma
  - Edmond, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Newton, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Spokane, Washington

REFERENCES:
- [Result] Staskin DR, Dmochowski RR, Sand PK, Macdiarmid SA, Caramelli KE, Thomas H, Hoel G. Efficacy and safety of oxybutynin chloride topical gel for overactive bladder: a randomized, double-blind, placebo controlled, multicenter study. J Urol. 2009 Apr;181(4):1764-72. doi: 10.1016/j.juro.2008.11.125. Epub 2009 Feb 23. PMID 19233423
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Drugs@FDA — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin Topical Gel: 1 g Oxybutynin topical gel
- Placebo Topical Gel: 1 g placebo topical gel
Period: Overall Study
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Started | 389 | 400
Completed | 346 | 355
Not Completed | 43 | 45
Not completed — Adverse Event | 19 | 13
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Lost to Follow-up | 9 | 8
Not completed — Physician Decision | 0 | 2
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel | Total
Number analyzed (Participants) | 389 | 400 | 789
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 246 | 260 | 506
  >=65 years | 143 | 140 | 283
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.50) | 59.3 (12.17) | 59.4 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 352 | 704
  Male | 37 | 48 | 85
Region of Enrollment [Number; unit: participants]
  United States | 389 | 400 | 789

OUTCOME MEASURES:

1. Primary Outcome: Baseline Average Number of Daily Incontinence Episodes
Description: Average number of daily incontinence episodes at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
Number of episodes | 5.4 (3.26) | 5.4 (3.28)

2. Secondary Outcome: Baseline Average Daily Urinary Frequency
Description: Number of daily urinary voids
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of urinary episodes
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
Number of urinary episodes | 12.4 (3.34) | 12.2 (3.32)

3. Secondary Outcome: Change From Baseline in Average Daily Urinary Frequency
Description: Change from baseline in average daily urinary frequency
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Number of urinary episodes
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
Number of urinary episodes | -2.7 (3.21) | -2.0 (2.82)

4. Primary Outcome: Change From Baseline in Average Daily Number of Incontinence Episodes
Description: Change from Baseline to Week 12 in average daily number of incontinence episodes
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Number of episodes
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
Number of episodes | -3.0 (2.73) | -2.5 (3.06)

5. Secondary Outcome: Baseline Average Urine Void Volume
Description: Baseline average urine void volume
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
mL | 163.4 (65.85) | 167.9 (68.40)

6. Secondary Outcome: Change From Baseline in Average Urine Void Volume
Description: Change from baseline to Week 12 in average urine void volume
Time Frame: Change from Baseline to Week 12
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Number analyzed (Participants) | 389 | 400
mL | 21.0 (65.33) | 3.8 (53.79)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Oxybutynin Topical Gel | Placebo Topical Gel
Serious Adverse Events (participants affected / at risk) | 7/389 | 10/400
Other Adverse Events (participants affected / at risk) | 176/389 | 145/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin Topical Gel (N=389) | Placebo Topical Gel (N=400)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Renal hemmorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin Topical Gel (N=389) | Placebo Topical Gel (N=400)
Application site pruritis (General disorders) | 8 (10) | 3 (3)
Bronchitis (Infections and infestations) | 9 (9) | 9 (11)
Constipation (Gastrointestinal disorders) | 7 (7) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 9 (11) | 13 (13)
Dizziness (Nervous system disorders) | 11 (12) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 29 (29) | 11 (12)
Fatigue (General disorders) | 8 (8) | 4 (4)
Gastroenteritis viral (Gastrointestinal disorders) | 8 (8) | 6 (6)
Headache (Nervous system disorders) | 19 (24) | 23 (28)
Nasopharyngitis (Infections and infestations) | 11 (11) | 9 (10)
Sinusitis (Infections and infestations) | 9 (10) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 21 (21) | 20 (20)
Urinary tract infection (Infections and infestations) | 27 (29) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less